CLINICAL TRIAL: NCT00082719
Title: Modulation of Death Effector Expression By Short-Term Exposure to Low-Dose Interferon
Brief Title: Short-Term Low-Dose Interferon Alfa in Treating Patients With Cancer of the Urothelium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0172; P50CA091846 (NIH); P30CA016672 (NIH); MDA-ID-030172 (Other: UT MD Anderson Cancer Center); CDR0000355831 (Registry Identifier: NCI PDQ); NCI-2012-02015 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Bladder Cancer; Urethral Cancer
Keywords: stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer; localized transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; metastatic transitional cell cancer of the renal pelvis and ureter; anterior urethral cancer; posterior urethral cancer; urethral cancer associated with invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Interferon-alpha; Interferon alpha-2; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Experimental): Low-dose interferon alfa subcutaneously (SC) twice daily.
  Interventions: Biological: Recombinant Interferon Alfa
- Arm II (Experimental): Interferon alfa as in arm I at a higher dose.
  Interventions: Biological: Recombinant Interferon Alfa
- Arm III (Experimental): Interferon alfa SC once daily.
  Interventions: Biological: Recombinant Interferon Alfa
- Arm IV (Experimental): Interferon alfa as in arm III at a higher dose.
  Interventions: Biological: Recombinant Interferon Alfa

INTERVENTIONS:
Biological: Recombinant Interferon Alfa — In all arms, treatment begins at pre-operative visit and continues until cystoscopy.
  Arm I: Low-dose interferon alfa subcutaneously (SC) twice daily. Arm II: Interferon alfa as in arm I at a higher dose. Arm III: Interferon alfa SC once daily. Arm IV: Interferon alfa as in arm III at a higher dose.
  Other Names: Interferon Alfa 2b; Intron A

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of tumor cells and slow the growth of urothelial cancer.

PURPOSE: This randomized phase I trial is studying how well low-dose interferon alfa works in treating patients with cancer of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the modulation of apoptosis-related pathways in patients with cancer of the urothelium treated with short-term low-dose interferon alfa.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 4 treatment arms.

In all arms, treatment begins at the time of the pre-operative visit and continues until the time of cystoscopy.

* Arm I: Patients receive low-dose interferon alfa subcutaneously (SC) twice daily.
* Arm II: Patients receive interferon alfa as in arm I at a higher dose.
* Arm III: Patients receive interferon alfa SC once daily.
* Arm IV: Patients receive interferon alfa as in arm III at a higher dose. In all arms, treatment continues in the absence of unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically proven urothelial cancer, known or suspected (e.g. by outside evaluation) to be muscle-invasive, and be scheduled for cystoscopy and transurethral biopsy as part of their routine evaluation at M. D. Anderson.
2. Patients must understand the investigational nature of this study and provide written, informed consent.

Exclusion Criteria:

1. Patients who are pregnant or lactating are not eligible. Women of child-bearing potential must have a negative pregnancy test before starting therapy.
2. Patients with current symptoms suggestive of clinically significant affective disorder.
3. Patients taking more than physiologic replacement doses of corticosteroids are not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Descriptive Data on Expression of Death Effectors in Context of Low-dose Interferon | 2 Years
  Data collection continues with treatment in absence of unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish M. Kamat, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org